CLINICAL TRIAL: NCT03349476
Title: Left Atrial Anatomy Reconstruction Using Model Based Fast Anatomical Mapping
Brief Title: Model Based Fast Anatomical Mapping
Acronym: MFAM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: study closed prior to meeting enrollment goal due to difficulty enrolling.
Sponsor: Vivek Reddy (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Vivek Reddy, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-02-329
Record Dates: First submitted 2017-11-17; First posted 2017-11-21 (Actual); Results first posted 2023-10-27 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Paroxysmal Atrial Fibrillation; Persistent Atrial Fibrillation
Keywords: Atrial Fibrillation; AFIB; Ablation; Paroxysmal; Persistent
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- MFAM (Experimental): The mFAM Workstation is a computerized system used to reconstruct the shape of the left atrium of the heart, by fitting a parametric shape model to points data acquired by a catheter.
  The mFAM Workstation uses recorded catheter positions and other data inputs collected from various types of multi-electrode catheters and generates output data files that can be displayed as a 3D anatomic structure.
  Interventions: Device: MFAM

INTERVENTIONS:
Device: MFAM — Specifically, the mFAM Workstation accesses stored data of recorded electronic heart activity that has been obtained by conventional electrophysiological methods, using multi-electrode catheters placed in the heart (data inputs) for collection. Using proprietary software algorithms, the mFAM Workstation analyzes these data inputs and generates 3D anatomical structure.
  mFAM improves on the FAM functionality by applying a model-based approach for reconstruction of left atrial chamber anatomy

SUMMARY:
This prospective, multicenter observational study will examine the ability of model based fast anatomical mapping (mFAM) to create left atrial (LA) geometry for atrial fibrillation ablation.

DETAILED DESCRIPTION:
This prospective, multicenter observational study will examine the ability of model based fast anatomical mapping (mFAM) to create left atrial (LA) geometry for atrial fibrillation ablation.

Specifically, the study will assess the following issues in atrial fibrillation ablation:

1. Accuracy of map (defined as the distance between the ablation points and the surface of the mFAM geometry)
2. Left atrial geometry creation time
3. Fluoroscopy time

The clinical team will hypothesize that this approach will lead to accurate LA geometry creation more rapidly and using less fluoroscopy than standard techniques

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Have AF as follows:

  1. Paroxysmal AF - defined as AF that is non-sustained (terminate without electrical or pharmacologic cardioversion) lasting < 7 days.
  2. Persistent AF - defined as AF that is sustained > 7 days. Episodes of AF which are terminated by electrical or pharmacologic cardioversion after ≥ 48 hours of AF, but prior to 7 days, should also be classified as persistent AF episodes.
* Are planned to undergo a first catheter ablation procedure (prior typical atrial flutter is allowed)
* Have the ability to understand the requirements of the study and sign the informed consent form.
* Are willing to adhere to study restrictions and comply with all post-procedural follow-up requirements

Exclusion Criteria:

* Rheumatic heart disease,
* Current intra-cardiac thrombus
* Class IV HF
* Unable to sign consent
* Unstable angina
* Recent cerebral ischemic events
* Contradiction to anticoagulation
* Prior cardiac surgery
* Complex congenital heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohit Turagam, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Vivek Reddy, MD, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- MFAM: The mFAM Workstation is a computerized system used to reconstruct the shape of the left atrium of the heart, by fitting a parametric shape model to points data acquired by a catheter.
  The mFAM Workstation uses recorded catheter positions and other data inputs collected from various types of multi-electrode catheters and generates output data files that can be displayed as a 3D anatomic structure.
  MFAM: Specifically, the mFAM Workstation accesses stored data of recorded electronic heart activity that has been obtained by conventional electrophysiological methods, using multi-electrode catheters placed in the heart (data inputs) for collection. Using proprietary software algorithms, the mFAM Workstation analyzes these data inputs and generates 3D anatomical structure.
  mFAM improves on the FAM functionality by applying a model-based approach for reconstruction of left atrial chamber anatomy
Period: Overall Study
Arm/Group | MFAM
Started | 109
Completed | 106
Not Completed | 3
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Arm/Group | MFAM
Number analyzed (Participants) | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.7 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 104
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 104
  More than one race | 0
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: mMap Scoring Questionnaire
Description: mMap Scoring Questionnaire: Tool used by operators to rate the accuracy of the map based on the distance between ablation points and accuracy of anatomy compared to the mapped mFam geometry.
  Total score from 1-7, with lower score indicating not representing (misleading) and higher score indicating agreement (accurate)
Time Frame: hospital discharge, average 24 hours post procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MFAM
Number analyzed (Participants) | 109
score on a scale | 5.3 (0.19)

2. Secondary Outcome: Left Atrial Geometry Creation Time
Description: The amount of time it takes to create the geometrical map using Carto and MFAM during the ablation procedure
Time Frame: during the procedure up to 60 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | MFAM
Number analyzed (Participants) | 109
minutes | 6.4 (0.25)

3. Secondary Outcome: Fluoroscopy Time
Description: Fluoroscopy (radiation) time for left atrial anatomy creation during the ablation procedure
Time Frame: hospital discharge, average 24 hours post procedure
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | MFAM
Number analyzed (Participants) | 109
seconds | 10.3 (33.5)

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | MFAM
All-Cause Mortality (participants affected / at risk) | 0/109
Serious Adverse Events (participants affected / at risk) | 1/109
Other Adverse Events (participants affected / at risk) | 2/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MFAM (N=109)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Right Lower Lobe Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MFAM (N=109)
Urinary Retention (Renal and urinary disorders) | 1
Recurrent Atrial Fibrillation (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/76/NCT03349476/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-23): https://cdn.clinicaltrials.gov/large-docs/76/NCT03349476/ICF_001.pdf